CLINICAL TRIAL: NCT02988284
Title: Investigating the Gait Variability in Healthy Individuals
Brief Title: Gait Variability in Healthy Youngs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, Research Assistant, PhD, PT, Hacettepe University
Other Study IDs: G01
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Gait variability

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
Three hundred healthy individuals will be participants of the study. Participants will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass, will be recorded. Gait parameters (step length, variation of step length) will evaluate with Gait trainer Biodex 2, at participant's preferred speed.

DETAILED DESCRIPTION:
Three hundred healthy individuals will be participants of the study. Participants will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass, year, side and level of limb loss will be recorded. Gait parameters (step length, variation of step length) will evaluate with Gait Trainer Biodex 2, at participant's preferred speed. To eliminate the learning effect, participants practiced at treadmill to determine appropriate gait speed. Once participants implied the preferred speed, they asked to walk at their self selected speed for 6 minutes. Data was recorded between the 4nd and 6th minutes at walk.

ELIGIBILITY:
Inclusion Criteria:

Want to participate

Exclusion Criteria:

Have passive joint limitation at extremities Surgery at last 5 year Systemic problems such as neurologic disorders, rheumatoid disorders… Another orthopedic anomalies

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Step length variability assesment while walking. | Initially evaluation at first minute

IPD SHARING:
Plan to Share IPD: Undecided